CLINICAL TRIAL: NCT04544150
Title: Gastrointestinal Manifestations in COVID-19: Symptoms and Signs and Its Impact on the Outcome
Brief Title: Gastrointestinal Manifestations Among Patients With COVID19
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Abu Elfatth, Al-rahji University Hospital, Faculty of Medicine, Assiut, Egypt, Assiut University
Other Study IDs: COVID19 and GUT
Record Dates: First submitted 2020-09-08; First posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:

SUMMARY:
many patients with confirmed infection with COVID-19 suffer from different symptoms and signs of gastrointestinal symptoms

DETAILED DESCRIPTION:
many patients with COVID1-9 infection experienced many intestinal symptoms mainly abdominal pain, vomiting, and diarrhea. This study aimed to assess the frequency of GIT manifestations among patients with COVID-19 and its impact on the outcome

ELIGIBILITY:
Inclusion Criteria:

* all patients with COVID19

Exclusion Criteria:

* patient refusal to participate in the study

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: all patients with COVID 19 infection
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
frequency of GIT symptoms among patients with COVID-19 infection | Baseline
  any GIT symptoms in such patients were recorded

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abu elfatth, Principal Investigator — Assuit University Hospitals
Locations (1):
- Ahmed, Al Minyā, Alminya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
to public
Supporting Information: Study Protocol
Time Frame: Baseline
URL: https://journals.sagepub.com/doi/full/10.1177/2050640620927955

REFERENCES:
- [Background] Peck-Radosavljevic M, Danese S, Hartmann D, Saftoiu A, Van Hootegem P; UEG Public Affairs Committee. COVID-19 and digestive health. United European Gastroenterol J. 2020 Jun;8(5):624-626. doi: 10.1177/2050640620927955. No abstract available. PMID 32450785